CLINICAL TRIAL: NCT06402890
Title: The Effect of Vitamin C-enriched Collagen Combined With Resistance Training on Muscle-tendon Unit Properties in Middle-aged Men and Women
Brief Title: Resistance Training and Hydrolyzed Collagen Supplementation in Middle-aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 300
Record Dates: First submitted 2024-04-17; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Diet; Food; Nutrition
Keywords: Hydrolyzed collagen; Middle-age; Resistance training; Tendon properties
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Before the intervention commenced, a laboratory technician (independent to the study) made up the dry ingestions all the 30 g doses of hydrolyzed collagen (HC), and calorie matched placebo and stored in sachets. These sachets were labelled as with the participants name. The technician randomly assigned either HC or placebo to participants who were pair matched (Excel 2016, Microsoft, Washington, USA). The groupings and contents of the sachets were unknown to the researcher and the participants, who all remained blinded until data collection and analysis were complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training with hydrolyzed collagen in health, active, middle-aged men (Experimental): Middle-aged, trained males completed 12-weeks of a supervised, progressive resistance training programme while consuming 30 g of hydrolyzed collagen or a calorie matched placebo beverage.
  Interventions: Dietary Supplement: Resistance training with collagen supplementation
- Resistance training with hydrolyzed collagen in healthy, active, middle-aged women (Experimental): Middle-aged, trained females completed 8-weeks of a supervised, progressive resistance training programme while consuming 30 g of hydrolyzed collagen or a calorie matched placebo beverage
  Interventions: Dietary Supplement: Resistance training with collagen supplementation

INTERVENTIONS:
Dietary Supplement: Resistance training with collagen supplementation — Participants performed 24 lower limb resistance training sessions over under supervision from the principal investigator. Participants were pair-matched, then allocated to hydrolysed collagen (COL) or a calorie-matched beverage comprising maltodextrin and non-caloric sweetener (PLA). Both COL and PLA consumed their respective supplements in conjunction with each resistance training session.
  Baseline assessments of strength were used to set initial training loads. An example of weekly training is included below for indicative purposes:
  Week 1 protocol:
  Day 1:
  * Barbell squat, 4 sets @ 90% 10-RM
  * Romanian deadlift, 4 sets @ 90% 10-RM
  Day 2:
  * Hex bar deadlift, 4 sets @ 90% 10-RM
  * Dumbbell goblet squat, 4 sets @ 90% 10-RM
  Linear progression adjusted weekly loads. If participants completed the prescribed sets and reps, loads increased by 2.5-5 % the following week.

SUMMARY:
The aim of this clinical trial is to investigate the longitudinal effects of hydrolyzed collagen ingestion combined with resistance training on muscle-tendon unit structure and function in middle-aged males and females.

The main research questions this clinical trial aims to answer are:

1. Does resistance training with hydrolyzed collagen ingestion lead to greater changes in tendon properties than resistance training alone in middle-aged health men and women?
2. Does resistance training with hydrolyzed collagen ingestion lead to greater changes in muscle size than resistance training alone?
3. Does resistance training with hydrolyzed collagen lead to greater increases in strength and power compared to resistance training alone in middle-aged, healthy men and women?

Participants will be randomly assigned to collagen or placebo groups. Participants will perform 24 sessions of high intensity resistance training across 12-weeks. Alongside each training session, participants will consume a beverage containing hydrolyzed collagen or maltodextrin, with both beverages containing vitamin C.

Researchers will compare the collagen and placebo groups to see if there would be beneficial effects on changes in muscle and tendon that are greater than resistance training alone. To achieve this, an dynamometry will be used to assess lower limb strength and ultrasound will be used to measure the morphological, mechanical, and material properties of the patellar tendon, as well the size and architecture of the vastus lateralis muscle.

DETAILED DESCRIPTION:
Healthy, active, middle-aged men and women will ingest a beverage containing 30 g of hydrolyzed collagen with 50 mg of vitamin C or a calorie matched beverage (maltodextrin), also with 50 mg of vitamin C combined with high-volume, high-intensity resistance training for the lower body on 2 - 3 occasions per week for 8-12 weeks.

The aim of this study was to investigate the effect of combining hydrolyzed collagen with resistance training in middle-aged men and women.If supplementation with hydrolyzed collagen leads to a greater change in tendon size, stiffness, and Young's modulus than resistance training alone, this will allow us to recommend this type of intervention to young athletes seeking to improve tendon health and/or athletic performance. This is the first study to investigate the combination of hydrolyzed collage supplementation with resistance training in middle-aged men and women. If supplementation with hydrolyzed leads to greater improvements in tendon size, stiffness, strength and/or power, this will allow us to recommend this type of intervention to middle-aged athletes/trainees seeking to improve tendon health, reduce injury risk, or enhance athletic performance.

The experimental design of both arms will be the same, however Arm 1 will be health, middle-aged male participants and Arm 2 will be health, middle-aged female participants.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active or competing in Masters sport
* No history of patellar tendon injuries in the past 6 months
* No history of lower limb musculoskeletal injuries in the past 6 months
* Non-smokers (including e-cigarettes)
* Free from cardiovascular and metabolic diseases

Exclusion Criteria:

* Age < 35 years or > 59 years
* Being vegan or vegetarian (due to the mammalian source of collagen)
* Injury history incompatible with lower body resistance training
* Consumption of nutritional supplementation that purportedly affects muscle-tendon adaptation or recovery (i.e. protein powder, vitamin C, collagen)
* BMI over 30 kg/m2

Ages: 35 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
m. vastus lateralis thickness (in millimetres) | 8-12 weeks' training and nutrition intervention
  Ultrasonography was used to determine changes in muscle thicknessprotocols
m. vastus lateralis fascicle pennation angle (in degrees) | 8-12 weeks' training and nutrition intervention
  Ultrasonography was used to determine the pennation angle of fascicles as they insert into the aponeurosis
Patellar tendon cross sectional area (in squared millimetres) at 3 regions along the tendon length | 8-12 weeks' training and nutrition intervention
  Ultrasonography was used to determine changes in tendon cross sectional area at 25, 50, and 75 % of tendon length
Patellar tendon stiffness (in Newtons per millimetre) | 8-12 weeks' training and nutrition intervention
  Synchronized ultrasonography, dynamometry, and surface electromyography were used to determine changes in patellar tendon stiffness
Bilateral vertical countermovement jump height (in centimetres) | 8-12 weeks' training and nutrition intervention
  Changes in jump height were estimated by use of the Optojump system (Microgate, Bolzano, Italy) and force plates (Force Decks Dual Force Plate System, VALD, Charlotte NC, USA).
Knee extensor maximal isometric torque (in Newton metres) | 8-12 weeks' training and nutrition intervention
  Changes in maximal knee extension strength were measured using isometric dynamometry (Biodex System 3, IPRS Mediquipe Limited, Lancashire, UK)
Knee extensor rate of torque development (in Newton metres per second) | 8-12 weeks' training and nutrition intervention
  Changes in explosive knee extension strength were measured using isometric dynamometry (Biodex System 3, IPRS Mediquipe Limited, Lancashire, UK)
Barbell back squat 10-repetition maximum (in kilograms) | 8-12 weeks' training and nutrition intervention
  Changes in dynamic lower body strength were measured using the maximum load during 10 repetitions of the barbell back squat exercise with standardised technique
Bilateral horizontal broad jump distance (in centimetres) | 8-12 weeks' training and nutrition intervention
  Changes in maximal horizontal displacement were measured as the maximum distance covered during a broad jump on standardised surface without footwear
Lower limb maximal isometric force (in Newtons) | 8-12 weeks' training and nutrition intervention
  Force plates (Force Decks Dual Force Plate System, VALD, Charlotte NC, USA) were used to measure changes in maximal multi-joint isometric strength during the mid-thigh pull exercise
Lower limb isometric rate of force development (in Newtons per second) | 8-12 weeks' training and nutrition intervention
  Force plates (Force Decks Dual Force Plate System, VALD, Charlotte NC, USA) were used to measure changes in explosive multi-joint isometric strength during the mid-thigh pull exercise
20-metre sprint time (in seconds) | 8-12 weeks' training and nutrition intervention
  Double photocell timing gates (Witty System, Microgate SRL, Bolzano, Italy) were used to measure changes in time taken to cover 20-metres during an all out sprint on a standardised surface

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Erskine, PhD, Study Director — Liverpool John Moores University; Christopher D Nulty, MSc, Principal Investigator — Liverpool John Moores University
Locations (1):
- Dr Rob Erskine, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT06402890/Prot_SAP_ICF_000.pdf